CLINICAL TRIAL: NCT00041262
Title: A Prospective Randomized Trial Comparing Standard Chemotherapy Followed By Resection Versus Infusional Chemotherapy In Patients With Resectable Adenocarcinoma Of The Oesophagus
Brief Title: Combination Chemotherapy in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: MRC-OE05; CDR0000069457 (Registry Identifier: PDQ (Physician Data Query)); EU-20204
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-03

CONDITIONS: Esophageal Cancer
Keywords: stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Epirubicin; Fluorouracil; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: epirubicin hydrochloride
Drug: fluorouracil
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective in treating esophageal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of combination chemotherapy in treating patients who are undergoing surgery for esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival and quality of life of patients with resectable adenocarcinoma of the esophagus treated prior to surgery with standard chemotherapy comprising cisplatin and fluorouracil versus prolonged infusional chemotherapy comprising cisplatin, epirubicin, and fluorouracil.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I (Standard chemotherapy): Patients receive cisplatin IV over 4 hours on days 1-4 and fluorouracil IV continuously on days 1-4. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (Infusional chemotherapy): Patients receive cisplatin IV over 4 hours on day 1, epirubicin IV on day 1, and fluorouracil IV continuously. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery 4-6 weeks after the last dose of fluorouracil in arm I or anytime after the fluorouracil infusion is completed in arm II.

Quality of life is assessed at baseline, immediately before starting the last course of chemotherapy, immediately before surgery, 6 weeks post-operatively, and at 6, 9, 12, 18, and 24 months after randomization.

Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: Approximately 1,300 patients (650 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the esophagus or type 1 or 2 tumors of the gastroesophageal junction

  * Stage IIB or greater by spiral or multi-slice CT scan and endoscopic ultrasound
  * Amenable to primary surgery with curative intent
* No para-aortic/celiac lymphadenopathy greater than 1 cm on CT scan and/or greater than 6 mm on endoscopic ultrasound
* No disease invading the airways, aorta, pericardium, or lung
* No liver, lung, or other distant metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Liver function tests no greater than 1.5 times normal

Renal:

* Glomerular filtration rate greater than 60 mL/min

Cardiovascular:

* Ejection fraction greater than 50% OR
* Normal echocardiograph

Pulmonary:

* FEV1 greater than 1.5 L

Other:

* Not pregnant or nursing
* No prior primary malignancy
* No significant medical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2004-11

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Disease-free survival
Local control
Morbidity from surgery and chemotherapy
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Derek Alderson, MD, Study Chair — University Hospital Birmingham
Locations (1):
- Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England, United Kingdom

REFERENCES:
- [Derived] Alderson D, Cunningham D, Nankivell M, Blazeby JM, Griffin SM, Crellin A, Grabsch HI, Langer R, Pritchard S, Okines A, Krysztopik R, Coxon F, Thompson J, Falk S, Robb C, Stenning S, Langley RE. Neoadjuvant cisplatin and fluorouracil versus epirubicin, cisplatin, and capecitabine followed by resection in patients with oesophageal adenocarcinoma (UK MRC OE05): an open-label, randomised phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1249-1260. doi: 10.1016/S1470-2045(17)30447-3. Epub 2017 Aug 4. PMID 28784312